CLINICAL TRIAL: NCT01285063
Title: Combined Physical Activity and Diet Intervention for the Treatment of Overweight and Obesity in Kindergarten Children
Brief Title: Intervention Study for Overweight and Obese Kindergarten Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not successful in raising money for this project
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mc01162010ctil
Record Dates: First submitted 2010-12-07; First posted 2011-01-27 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Overweight; Obesity; Physical Fitness
Keywords: overweight; obesity; physical fitness; kinder garden; preschool
MeSH Terms: conditions — Overweight; Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- physical activiy & nutrition (Experimental): 25 kindergarten children in the ages of 4-6 who defined as suffering from overweigh (BMI percentage 85-95) or obesity (above BMI percentage 95).
  Non-generalization criteria: children who suffer from obesity due to organic disease or children who take medicine which may influence body weight (e.g., steroids) will be excluded from the research.
  Interventions: Other: Multidisciplinary intervention: physical activity, dietary instructions and behavioral treatment.

INTERVENTIONS:
Other: Multidisciplinary intervention: physical activity, dietary instructions and behavioral treatment. — 3 months intervention. Nutritious plan: includes 6 meetings of the child and his or her parents with a dietician from the center.
  Physical activity: physical trainings of 60 minutes each will be held twice a week.
  behavioral treatment: all the participants will take part it a 45 minutes meeting of movement therapy once a week. The goal of such meeting is to strengthen nutritious and physical activity habits and to assimilate positive change in the participants' lifestyle.

SUMMARY:
The goal of the this study is to create an interdisciplinary program which includes intervention in the fields of nutrition, physical activity and behavior in order to treat obesity and overweight among kindergarten children and to examine the influence of such program on the BMI,BMI%, physical fitness, knowledge and preferences in the said fields among the participants.

DETAILED DESCRIPTION:
Subjects, goals and objective:

Obesity is the most common chronic children disease of the modern era. The number of children who suffer from obesity is increasing to scales of epidemic. The frequency of obesity among kindergarten children (ages of 2-5) in the United States is approximately 14%, whereas among children of those ages in the center of Israel there is a risk of 25% to obesity and overweight.

Obesity is not only a cosmetic problem but also constitutes the #1 risk factor for common medical problems, such as: hyperlipidemia, high blood pressure, glucose intolerance, type 2 diabetes, arteriosclerosis, asthma, orthopaedic problems and psychological problems. A comprehensive review that was recently published showed that among fat children, intensive intervention programs which include nutrition consulting, physical training and behavioral change are the most effective to treat obesity.

Children who suffer from obesity have a greater risk to become fat adults and the older the child the greater the risk becomes. Therefore, it is highly important to treat such obesity in the youngest age possible. Moreover, along with the change of nutritious preferences, a great emphasize should be given to physical activity in order to reduce the BMI percentage and improve the physical fitness.

The goal of the paper is to create an interdisciplinary program which includes intervention in the fields of nutrition, physical activity and behavior in order to treat obesity and overweight among kindergarten children and to examine the influence of such program on the BMI,%BMI, physical fitness, knowledge and preferences in the said fields among the participants.

Place: The intervention program will be held in the sports and health center for children and youth at "Meir" medical center.

The intervention group: 25 kindergarten children in the ages of 4-6 who defined as suffering from overweigh (BMI percentage 85-95) or obesity (above BMI percentage 95).

Non-generalization criteria: children who suffer from obesity due to organic disease or children who take medicine which may influence body weight (e.g., steroids) will be excluded from the research.

The control group: 25 kindergarten children in similar ages who defined as suffering from overweigh (BMI percentage 85-95) or obesity (above BMI percentage 95) and who do not participate in any intervention program.

The research plan Nutritious plan: includes 6 personal meetings, 30-45 minutes each, of the child and his parents with a dietician from the center. The meetings will include nutritious evaluation and will focus on nutritious education.

Physical activity: physical trainings of 45 minutes each will be held twice a week and be guided by a qualified trainer. In order to encourage the participants to take responsibility for the process, the children will be asked to further practice during the weeks and conduct little assignments which will be given by the trainer.

Additionally, all the participants will take part it a 45 minutes meeting of movement therapy once a week. Such meeting will be held by a qualified trainer. The goal of such meeting is to strengthen nutritious and physical activity habits and to assimilate positive change in the participants' lifestyle.

Evaluation index: height, weight, BMI and BMI percentage,"nutrition and physical activity knowledge and preferences" questionnaire. The questionnaire is an instrument to evaluate the knowledge and preferences of children in the ages of 4-8 in the fields of nutrition and physical activity.

Evaluation of physical fitness: "back and forth" running test for a 10m distance.

ELIGIBILITY:
Inclusion Criteria:

* children in ages of 4-6 who defined as suffering from overweigh (BMI percentage 85-95) or obesity (above BMI percentage 95).

Exclusion Criteria:

* children who suffer from obesity due to organic disease or children who take medicine which may influence body weight (e.g., steroids) will be excluded from the research.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
reduction of the BMI percentage among the participants in comparison to the control group. | every 2 weeks.
  height, weight, BMI and BMI percentage will be documented after each meeting with the dietitian.

SECONDARY OUTCOMES:
Improvement in the physical fitness of the participants in comparison to the control group. | Day 1 and after 3 months.
  "Back and forth" running test for a 10m distance.
Positive change in the knowledge and preferences of the participants in the fields of nutrition and physical activity in comparison to the control group. | Day 1 and after 3 months.
  "Nutrition and physical activity knowledge and preferences" questionnaire. The questionnaire is an instrument to evaluate the knowledge and preferences of children in the ages of 4-8 in the fields of nutrition and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Tali Sinai, Dr, Study Chair — The hebrew university, Jerusalem
Locations (1):
- the sports and health center for children and youth at "Meir" medical center, Kfar Saba, Israel